CLINICAL TRIAL: NCT01071460
Title: The FlexStent-Registry, Evaluation of Efficacy and Safety of the FlexStent Femoropopliteal Self-Expanding Stent System
Brief Title: Evaluation of Efficacy and Safety of the FlexStent Self-Expanding Stent System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Provascular GmbH (Other)
Responsible Party: Dierk Scheinert, MD, Park Krankenhaus Leipzig
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prov 01-2009; 147-2009-06072009 (Other: Ethic Committee at the University of Leipzig, Germany)
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Efficacy of the Study Device
Keywords: PAD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SFA Stenting (Other)
  Interventions: Device: FlexStent Femoropopliteal Self-Expanding Stent System

INTERVENTIONS:
Device: FlexStent Femoropopliteal Self-Expanding Stent System — Peri-procedural management will be no different to routine SFA/Popliteal Artery intervention Standard medical therapy
  Procedural techniques will be identical to routine protocols for SFA/Popliteal Artery stenting. technique suggested:
  * Contralateral retrograde common femoral cross-over access or antegrade access
  * Target lower limb arteries fully imaged angiogram. with measurement of SFA/Popliteal Artery target lesion length and normal vessel diameter immediately above and below target lesion
  * Pre-stenting balloon dilatation of target lesion in all total occlusions and critical stenosis
  * Deployment of an appropriately sized FlexStent® to cover target lesion
  * Post-stent balloon dilate stent using a semi-compliant angioplasty balloon to enable accurate post-dilatation of stent to target diameter
  * Post stenting angiography assessing target lesion parameters, run-off vessel patency and complications

SUMMARY:
Purpose of this registry is to determine the efficacy and safety of the self-expanding, extra flexible FlexStent in patient with superficial femor/popliteal artery disease.

The stent has been developed to cope with the extreme requirements of the femoral artery/knee artery and is approved for usage at humans (EC-certified). It is designed to treat narrows of the femoral- and knee artery.

100 patients at 5 German hospital shall be enrolled. After stent implantation follow-up visits at 6 and 12 month take place.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) represents a major challenge to physicians in treating the Superficial Femoral (SFA) and Popliteal arteries. These arteries represent a harsh environment for any endovascular device. This disease is characterized by long occlusions with relatively low flow and with the vessels exposed to enormous mechanical stress. During flexing of the knee, the SFA/Popliteal arteries can bend, rotate, elongate and compress dramatically. An ideal stent designed for use in the SFA/Popliteal arteries would offer great ranges of movement while adequately supporting the arteries.

The FlexStent® stent provides a great range of motions for a highly flexible femoral artery while adequately supporting the vessel. The intended use for the FlexStent® stent is for the treatment of symptomatic femoropopliteal disease, primarily for atherosclerotic de novo native superficial femoral artery lesions.

The intent of this clinical registry is to demonstrate the efficacy and safety of the FlexStent® stent in patients with superficial femoral/ popliteal artery disease.

Hypothesis: the FlexStent® will be safe and efficacious in treating SFA/popliteal artery diseases.

Primary object: evaluation of efficacy of the FlexStent® measured by the in-stent restenosis using DUS following treatment, 6 and 12 MFU visits.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, male or female, must be between the ages of 35 to 85 years inclusive at the time of consent. A female of childbearing potential may be enrolled, provided she has a negative pregnancy test at Screening.
* Subjects must give written informed consent prior to participation in the study and must understand the purpose of this study and be willing to adhere to the study procedures described in this protocol.
* Rutherford Classification Category 2-4
* Single de novo lesion in the superficial femoro/popliteal artery
* Disease segment length ≤150mm

  ->70% diameter stenosis and occlusion
* Patent ipsilateral iliac artery
* Patent ipsilateral popliteal artery and at least 1 patent tibial artery in continuity to ankle
* Target reference vessel diameter 3.5-7.5 mm

Exclusion Criteria:

* Target lesion previously treated with a stent or surgery.
* Rutherford Classification Category 0,1,5 or 6.
* Inability to tolerate antithrombotic or antiplatelet therapies.
* Pregnancy.
* Other comorbidity risks which in the opinion of the investigator limit longevity or likelihood of complying with protocol follow up.
* Serum creatinine > 2.5 mg/dL.
* Myocardial infarction or stroke within 90 days of enrollment.
* Hypercoagulable state.
* Uncontrollable hypertension.
* Patients currently enrolled in any other clinical trial(s).

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
in-stent binary restenosis using DUS | after treatment, at 6 and 12 MFU

SECONDARY OUTCOMES:
technical success, defined as the ability to implant the stent with a residual angiographic stenosis no greater than 30% | at 6 and 12 MFU

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, Professor, Principal Investigator — Park-Krankenhaus Leipzig
Locations (3):
- Germany (3):
  - Herz-Zentrum Bad Krozingen Abteilung Angiologie, Bad Krozingen
  - Jüdisches Krankenhaus Berlin, Gefäßzentrum, Berlin
  - Park-Krankenhaus Leipzig, Leipzig